CLINICAL TRIAL: NCT05385497
Title: Combining Aerobic Exercise and Virtual Reality for Cognitive-motor Rehabilitation in Parkinson's Disease
Brief Title: Combining Aerobic Exercise and Virtual Reality for Cognitive-motor Rehabilitation in PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Texas Physical Therapy Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSC20220064H
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Parkinson's Disease
Keywords: Aerobic Exercise; Virtual Reality
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study will utilize a single group, pre-post design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined Aerobic Exercise (AE) and Virtual Reality (VR)-based program (Experimental): Individuals diagnosed with PD will participate in AE and VR.
  Interventions: Other: Aerobic Exercise; Device: Virtual Reality

INTERVENTIONS:
Other: Aerobic Exercise — Participants will perform a 30-minute exercise protocol (5 minutes warm-up and cool-down each and 20 minutes moderate intensity exercise) on a StepOne™ recumbent stepper
Device: Virtual Reality — Participants will interact with the virtual environment and view the gaming environment on a flat-screen TV placed in front of them at a suitable distance. The participants will play four games (50 repetitions/game divided into three blocks with 1-2 minutes rest between blocks), with the order of the games randomized in every session.

SUMMARY:
This project will provide preliminary data on the feasibility and effects of exercise and VR on motor behavior and neuroplasticity in PD. Results from this work will provide insight into whether combination interventions utilizing AE and VR have parallel effects on cognition, gait, and neuroplasticity in PD.

DETAILED DESCRIPTION:
In this pilot proof-of-concept study, the study team will recruit 10 individuals with Parkinson's disease who will perform aerobic exercise (AE) followed by virtual reality (VR). The study team will measure the effects of the intervention on dual task performance, clinical measures of gait, cognition, TMS measures and questionnaires pertaining to quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic PD (ages 18 - 85) in Hoehn and Yahr stages 1 - 3.
2. Subjects need to demonstrate a score of equal to or greater than 23 on the Mini Mental State Examination.

Exclusion Criteria:

1. Subjects with a history of other neurological diseases (i.e. stroke, multiple sclerosis).
2. Subjects with a history of severe cardiopulmonary disease, uncontrolled hypertension, orthostatic hypotension, uncontrolled diabetes, severe osteoporosis.
3. Subjects with a history of PD-specific surgical procedure such as deep brain stimulation etc.
4. Subjects with a history of head injury.
5. Subjects with a history of seizures or epilepsy,
6. Subjects who are currently pregnant
7. Subjects who use of medications that could alter corticomotor excitability or increase risk of seizure
8. Subjects with skull abnormalities, fractures, unexplained, recurring headaches.
9. Subjects who have cognitive or communication impairment that would affect participation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Gait speed | Baseline to 3 weeks
  10 Meter Walk Test for comfortable and fast gait speed (m/s).
Spatiotemporal Parameters | Baseline to 3 weeks
  Spatiotemporal measures of gait will be acquired with a gait mat during single and dual task conditions. Participants will perform 2 trials each at their self-selected speed for the single task and dual task conditions for the the gait tests.
Cognition | Baseline to 3 weeks
  Parkinson's disease (PD)-cognitive rating scale
Balance | Baseline to 3 weeks
  Balance will be tested with the Mini-BESTest (Balance Evaluation Systems Test), involving 14 different tasks to assess static and dynamic balance. The Mini-BESTest is a clinical test for the construct of dynamic balance. It consists of 14 items, divided into four subcomponents: anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait. Items are scored from 0 (unable or requiring help) to 2 (normal) on an ordinal scale, with the maximal total score of 28 points. A higher score indicates better balance.
Corticomotor excitability | Baseline to 3 weeks
  Change in Corticomotor excitability as measured with transcranial magnetic stimulation (TMS).

SECONDARY OUTCOMES:
Quality of Life Survey | Baseline to 3 weeks
  Change in QoL as assessed by PDQ-8, a self-reported Parkinson's Disease Questionnaire using 8 questions with the answers: Never, occasionally, sometimes, often or always (or cannot do at all). Scores range from 0-32 with a higher score indicating worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Sivaramakrishnan, PT, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- UT Health San Antonio- Dept. of Physical Therapy, San Antonio, Texas, United States